CLINICAL TRIAL: NCT05435729
Title: A Pharmacodynamics and Safety Study of DSP-9632P in Patients With Levodopa-Induced Dyskinesia in Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DD701105; jRCT2031220051 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2022-06-13; First posted 2022-06-28 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Levodopa-induced Dyskinesia; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Periods 1 and 2 in Part B will be conducted in a double-blinded manner. The subjects, all study staff including the investigator, drug concentration-measuring facility, drug residual amount-measuring facility, safety review team, and the Sponsor are kept blinded to the assignment of treatment during the period from the initiation of the study to database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DSP-9632P 27.5 mg in Periods 3 of Part A (Experimental): Single dose of DSP-9632P 27.5 mg in patients with levodopa-induced dyskinesia in Parkinson's disease
  Interventions: Drug: DSP-9632P 27.5 mg; Drug: Levodopa formulation
- DSP-9632P 82.5 mg in Periods 4 of Part A (Experimental): Single dose of DSP-9632P 82.5 mg in patients with levodopa-induced dyskinesia in Parkinson's disease
  Interventions: Drug: DSP-9632P 82.5 mg; Drug: Levodopa formulation
- DSP-9632P 55.0 mg in Period 1 or 2 of Part B (Experimental): Multiple dose of DSP-9632P 55.0 mg in patients with levodopa-induced dyskinesia in Parkinson's disease
  Interventions: Drug: Placebo; Drug: DSP-9632P 55.0 mg; Drug: Levodopa formulation

INTERVENTIONS:
Drug: DSP-9632P 27.5 mg — Single dose of DSP-9632P 27.5 mg
  Arms: DSP-9632P 27.5 mg in Periods 3 of Part A
Drug: DSP-9632P 82.5 mg — Single dose of DSP-9632P 82.5 mg
  Arms: DSP-9632P 82.5 mg in Periods 4 of Part A
Drug: Placebo — Placebo for DSP-9632P
  Arms: DSP-9632P 55.0 mg in Period 1 or 2 of Part B
Drug: DSP-9632P 55.0 mg — Multiple dose of DSP-9632P 55.0 mg
  Arms: DSP-9632P 55.0 mg in Period 1 or 2 of Part B
Drug: Levodopa formulation — Single dose of Levodopa formulation

SUMMARY:
This study is an open-label of single transdermal dose of DSP-9632P to evaluate the dopamine release derived from levodopa in brain, and a randomized, double-blind, placebo-controlled, 2-way crossover of multiple transdermal doses of DSP-9632P to evaluate the safety and tolerability in patients with levodopa-induced dyskinesia in Parkinson's disease.

DETAILED DESCRIPTION:
This study consists of Part A and Part B. Part A is an open-label part to evaluate the amount of striatal dopamine release derived from levodopa following single transdermal administration of DSP-9632P using 11Craclopride PET in patients with levodopa-induced dyskinesia in Parkinson's disease. Part A consists of screening, Period 1, Period 2, Period 3, Period 4, and follow-up period. Each period consists of 2 days, Day 1 and Day 2. There will be a 7-day or longer washout of DSP-9632P between Periods 3 and 4. Subjects will be hospitalized in each period.

Part B is a randomized, double-blind, placebo-controlled, crossover part to evaluate the safety and tolerability of DSP-9632P following multiple transdermal administration in patients with levodopa-induced dyskinesia in Parkinson's disease. Part B consists of screening, placebo lead-in period, baseline period, Period 1, Period 2, and follow-up period. Period 1 and Period 2 consist of 9 days. Subjects will be hospitalized for 10 days 9 nights from baseline period to Period 1 and for 9 days 8 nights in Period 2. There will be a 7-day or longer washout of DSP-9632P between Periods 1 and 2.

Subjects will concomitantly use any of the levodopa formulation from the time of informed consent to the end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject whose age is ≥ 50 and < 80 years at the time of informed consent.
2. Subject who is fully informed and understands the objectives, procedures, anticipated drug effects/pharmacological action and risks of the study and who voluntarily provides written consent to participate in the study.
3. Subject who has clinically established Parkinson's disease diagnosed by MDS clinical diagnostic criteria for Parkinson's disease (2015).
4. Subject who has a response to levodopa at screening in the opinion of the investigator.
5. Subject who is confirmed to have dopaminergic denervation with a specific binding ratio in the striatum, obtained by dopamine transporter SPECT (123I-FP-CIT, DAT scan®) performed prior to the study or at screening, that is lower than the lower limit of 95% confidence interval of healthy adults.
6. Subject who has a Hoehn & Yahr stage ≤ III in the ON state at screening.
7. Subject who has MDS-UPDRS Part IV-1 ≥ 2 and Part IV-2 ≥ 2 at screening.
8. Subject who is on treatment with levodopa formulation at least 3 times daily at screening.
9. Subject who is able to receive 11C-raclopride PET scans (Part A only).
10. Subject who has a score of ≥ 2 in any of questions of UDysRS Part 1B at screening (Part B only).
11. Subjects who can wear the glasses-type wearable device and agree to wear it (Part B only).
12. Subject who is able to comply with the study requirements, including physical examination, assessments, and reporting symptoms.
13. Subject who is willing to practice abstinence or use appropriate contraception as part of the subject's lifestyle from signing informed consent through 30 days after the last dose of study drug.
14. Subject who is on treatment with levodopa formulation at least 3 times daily and is treated with levodopa formulation with a fixed dosing regimen for at least 28 days prior to Period 1 (Part A) or prior to admission (Part B).
15. Subject who is in the ON state with dyskinesia every day for at least 30 minutes twice or more daily based on the PD home diary during the placebo lead-in period (Part B only).

Exclusion Criteria:

1. Subject with a clinically significant history of cardiovascular, hepatic, renal, endocrine, gastrointestinal, hematological, respiratory, or neurologic disease other than Parkinson's disease, determined by the investigator.
2. Subject who has a disorder or history of a condition that may interfere with drug metabolism or excretion including clinically significant abnormality of the hepatic or renal systems.
3. Subject with a history of epilepsy, convulsions, unexplained syncope or other unexplained loss of consciousness (except a single incident), or head trauma with loss of consciousness lasting more than 5 minutes.
4. Subject with a clinically significant abnormal 12-lead ECG or a screening 12-lead ECG for safety assessment that demonstrates any one of the following:

   1. Heart rate > 100 bpm or < 50 bpm
   2. QRS interval > 120 msec
   3. QTcF > 450 msec (male) or > 470 msec (female)
   4. PR interval > 200 msec
5. Subject with dermatosis or skin abnormality (eg, dermatitis, eczema, or dyschromatosis) at application sites.
6. Subject with a history of drug allergy or skin allergy.
7. Subject with a known sensitivity to any transdermal patch.
8. Subject with a history of drug abuse or narcotic abuse, or a positive urine drug screening at screening.
9. Subject who has a positive immunology at screening.
10. Subject with any clinically significant abnormal clinical laboratory value (hematology test, serum chemistry test, urinalysis, coagulation test, or lipid test) determined by the investigator at screening.
11. Subject with a history of biphasic dyskinesia, myoclonus, or apathy.
12. Subject with a current or history of psychiatric illness (eg, schizophrenia, bipolar disorder, depression) based on the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5).
13. Subject with Mini-Mental State Examination (MMSE) score of ≤ 23 at screening.
14. Subject who has received surgical therapy related to Parkinson's disease.
15. Subject who has previously received levodopa-carbidopa intestinal gel.
16. Subject who has previously received DSP-9632P.
17. Subject who has participated in any clinical study and received any investigational drug during the 90 days prior to screening visit, or who is currently participating in another clinical trial.
18. Subject who has experienced significant blood loss or donated blood (≥ 400 mL) during the 90 days prior to screening or donated 200 mL of blood or more during the 30 days prior to screening; has donated blood components during the 14 days prior to screening or intends to donate blood components or blood during the 30 days after the last study visit.
19. Subject who is in the opinion of the investigator unsuitable in any other way to participate in this study.
20. Subject who has a positive urine drug screening at admission.
21. Subject who has consumed caffein or smoked in 2 days prior to the admission or has consumed alcohol in 1 day prior to the admission (Part A only).
22. Subject who answers "yes" to "Suicidal Ideation" Items 4 or 5 on the C-SSRS at admission.
23. Subject who has used dopamine receptor antagonists (antipsychotics, metoclopramide, domperidone) within 14 days prior to Period 1.
24. Subject who has used serotonergic 5-HT1A/1B agonists/antagonists (tandospirone, sumatriptan, zolmitriptan, eletriptan, rizatriptan, naratriptan, Yokukansan) during the 14 days prior to Period 1.
25. Subject who has used therapeutic agents (monoamine oxidase B [MAO-B] inhibitors, zonisamide, istradefylline, anticholinergics) for Parkinson's disease other than levodopa formulations, dopamine receptor agonists and COMT inhibitors within 28 days prior to Period 1.
26. Subject who has used amantadine hydrochloride during the 28 days prior to Period 1.
27. Subject who has used antidepressants (tricyclic antidepressants, tetracyclic antidepressants, selective serotonin reuptake inhibitors [SSRI], serotonin/norepinephrine reuptake inhibitors [SNRI], or noradrenergic and specific serotonergic antidepressants [NaSSA], etc.) during the 28 days prior to Period 1.
28. Subject with a positive severe acute respiratory syndrome coronavirus 2 (SARSCoV-2) nucleic acid amplification test to be performed between screening and admission in Period 1, or clinical symptoms suggestive of infection with SARSCoV-2 before admission.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Binding potential of 11C-raclopride and Dopamine D2 receptor occupancy by Positron Emission Tomography (PET) in Part A | 1 day
  Evaluate the amount of striatal dopamine release derived from levodopa following single transdermal administration of DSP-9632P using 11C-raclopride PET in patients with levodopa-induced dyskinesia in Parkinson's disease
Incidence of adverse events (AEs), serious adverse events (SAEs), and AEs leading to treatment discontinuation in Part B | 7 days
  Evaluate the Incidence of AEs, SAEs, and AEs leading to treatment discontinuation of DSP-9632P following multiple once-daily transdermal administration for 7 days in patients with levodopa-induced dyskinesia in Parkinson's disease transdermal administration for 7 days in patients with levodopa-induced dyskinesia in Parkinson's disease

SECONDARY OUTCOMES:
Change from baseline in Unified Dyskinesia Rating Scale (UDysRS) score in Part A | 1 days
  Evaluate the change from baseline in UDysRS score following single transdermal administration of DSP-9632P in patients with levodopa-induced dyskinesia in Parkinson's disease
Change from baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score in Part A | 1 days
  Evaluate the change from baseline in MDS-UPDRS score following single transdermal administration of DSP-9632P in patients with levodopa-induced dyskinesia in Parkinson's disease
Incidence of adverse events (AEs), serious adverse events (SAEs), and AEs leading to treatment discontinuation in Part A | 1 days
  Evaluate the Incidence of adverse events (AEs), serious adverse events (SAEs), and AEs leading to treatment discontinuation of DSP-9632P following single transdermal administration in patients with levodopa-induced dyskinesia in Parkinson's disease
Cmax of levodopa in Part A | 1 days
  Evaluate the Cmax of levodopa following oral administration of levodopa formulation in patients with levodopa-induced dyskinesia in Parkinson's disease
Time of occurrence of Cmax (tmax) of levodopa in Part A | 1 days
  Evaluate the tmax of levodopa following oral administration of levodopa formulation in patients with levodopa-induced dyskinesia in Parkinson's disease
Area under the plasma concentration-time curve (AUC) of levodopa in Part A | 1 days
  Evaluate the AUC of levodopa following oral administration of levodopa formulation in patients with levodopa-induced dyskinesia in Parkinson's disease
Terminal elimination half-life (t1/2) of levodopa in Part A | 1 days
  Evaluate the t1/2 of levodopa following oral administration of levodopa formulation in patients with levodopa-induced dyskinesia in Parkinson's disease
Summary statistics of plasma concentrations of tandospirone and its metabolite 1-(2-Pyrimidyl) piperazine (1-PP) in Part A | 1 days
  Evaluate the summary statistics of plasma concentrations of tandospirone and 1-PP following single transdermal administration of DSP-9632P in patients with levodopa-induced dyskinesia in Parkinson's disease
Sum and maximum of change from baseline in UDysRS score in Part B | 7 days
  Evaluate the sum and muximum of change from baseline in UDysRS score following multiple once-daily transdermal administration of DSP-9632P for 7 days in patients with levodopa-induced dyskinesia in Parkinson's disease
Sum and maximum of change from baseline from MDS-UPDRS score in Part B | 7 days
  Evaluate the sum of change from baseline in MDS-UPDRS score following multiple once-daily transdermal administration of DSP-9632P for 7 days in patients with levodopa-induced dyskinesia in Parkinson's disease
Cmax of levodopa in Part B | 7 days
  Evaluate the Cmax of levodopa following oral administration of levodopa formulation in patients with levodopa-induced dyskinesia in Parkinson's disease
tmax of levodopa in Part B | 7 days
  Evaluate the tmax of levodopa following oral administration of levodopa formulation in patients with levodopa-induced dyskinesia in Parkinson's disease
AUC of levodopa in Part B | 7 days
  Evaluate the AUC of levodopa following oral administration of levodopa formulation in patients with levodopa-induced dyskinesia in Parkinson's disease
t1/2 of levodopa in Part B | 7 days
  with levodopa-induced dyskinesia in Parkinson's disease
Summary statistics of Plasma concentrations of tandospirone and 1-PP in Part B | 7 days
  Evaluate the Summary statistics of plasma concentrations of tandospirone and 1-PP following multiple once-daily transdermal administration of DSP-9632P for 7 days in patients with levodopa-induced dyskinesia in Parkinson's disease

OTHER OUTCOMES:
Absolute value and change from baseline in EuroQol 5 dimensions 5-level (EQ-5D-5L) total score in Part B | 7 days
  Evaluate the absolute value and change from baseline in EQ-5D-5L total score following multiple once-daily transdermal administration of DSP-9632P for 7 days in patients with levodopa-induced dyskinesia in Parkinson's disease
Absolute value and change from baseline in Parkinson's Disease Questionnaire-39 (PDQ-39) total score, score of 8 domains, and summary index score in Part B | 7 days
  Evaluate the absolute value and change from baseline in PDQ-39 total score, score of 8 domains, and summary index score following multiple once-daily transdermal administration of DSP-9632P for 7 days in patients with levodopa-induced dyskinesia in Parkinson's disease
Change from baseline in eye movement parameters (e.g. eye-blink rates) in Part B | 7 days
  Evaluate the eye movement parameters (eg, eye-blinking rates) following oral administration of levodopa formulation and transdermal administration of DSP-9632P in patients with levodopa-induced dyskinesia in Parkinson's disease

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Medical School Hospital, Bunkyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No